CLINICAL TRIAL: NCT03219541
Title: Feasibility and Acceptability of a Text Messaging Intervention to Increase Smoking Cessation in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00630
Record Dates: First submitted 2017-07-06; First posted 2017-07-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Automated mobile phone text (Active Comparator): Subjects will receive 2 messages per day in the pre-quit phase, 3 messages per day on the quit date and the first week in the post-quit phase, and 2 messages per day in the last 3 weeks of the intervention. During the intervention, participants will receive a text question at the end of every day asking you "How many cigarettes have you smoked today?"
  Interventions: Behavioral: Interventional Automated mobile phone text
- Control Texts (Placebo Comparator): The intervention will consist of a 3-day pre-quit period and then a 4-week post-quit period. Participants will receive 2 text questions each week asking the number of smoking days in the past week and the average number of cigarette smoked per day.
  Interventions: Behavioral: Control Automated mobile phone text

INTERVENTIONS:
Behavioral: Interventional Automated mobile phone text — Participants will receive 2 messages per day in the pre-quit phase, 3 messages per day on the quit date and the first week in the post-quit phase, and 2 messages per day in the last 3 weeks of the intervention.
  Arms: Interventional Automated mobile phone text
Behavioral: Control Automated mobile phone text — Participants will receive 2 text questions each week asking the number of smoking days in the past week and the average number of cigarette smoked per day.
  Arms: Control Texts

SUMMARY:
The purpose of this study is to develop and then test the feasibility, acceptability, and preliminary effect of a bidirectional text message smoking cessation intervention among Vietnamese smokers in Hanoi, Vietnam. The specific aim are: 1) To develop a smoking cessation text message library among Vietnamese smokers; 2) To evaluate message preferences, and the feasibility and acceptability of the bidirectional text message smoking cessation intervention; and 3) To assess the preliminary effect of a bidirectional mobile phone text message intervention on biochemically validated smoking abstinence.

DETAILED DESCRIPTION:
For two-arm randomized control (RCT) pilot study (AIM 3), 100 current smokers will be observed to examine the preliminary effect of bidirectional SMS smoking cessation intervention. Subjects will be randomized into two groups (intervention vs. control), and compare the carbon monoxide (CO) validated 7-day point prevalence smoking abstinence rates at 4-week follow-up between intervention group (SMS smoking cessation treatment) and control group (assessment texts only).

Investigators will administer surveys at baseline, 4- and 12-weeks, and assess daily cigarette consumption using text message surveys. After the intervention, they will randomly select 10 participants from the intervention group to attend semi-structured interviews to obtain more in-depth understanding about the usefulness, usability, and acceptability of the intervention. Findings from the pilot RCT will be used to derive an estimate of the effect size, power, and sample size for a full-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* smoke ≥10 cigarettes per day
* capability to read and communicate
* plan to quit in the next 30 days
* has a mobile phone
* has experience using mobile phone text messaging during the past 6 months.

Exclusion Criteria:

* Under smoking cessation treatment or is participating in other tobacco cessation intervention
* pregnant or breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | 12 Weeks
  Measured by ranking the mean score of each message

SECONDARY OUTCOMES:
Number of quit attempts | 12 Weeks
  Measured using the 12-item Cigarette Dependence Scale (CDS)
Percentage of respondents who have made at least one quit attempt during the intervention period, | 12 Weeks
  Measured using the Smoking Absitinence Questionnaire (SAQ)
Percent decrease in cigarette consumption per day at 2- and 4-week follow-ups compared to baseline | 4 Weeks
  Measured using the Smoking Absitinence Questionnaire (SAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Jiang N, Nguyen N, Siman N, Cleland CM, Nguyen T, Doan HT, Abroms LC, Shelley DR. Adaptation and Assessment of a Text Messaging Smoking Cessation Intervention in Vietnam: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Oct 8;9(10):e27478. doi: 10.2196/27478. PMID 34623318